CLINICAL TRIAL: NCT02623049
Title: Direct Oral Anticoagulants Pharmacodynamics in Octogenarian Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, shmuel fuchs, Professor, Rabin Medical Center
Other Study IDs: 0590-15
Record Dates: First submitted 2015-11-19; First posted 2015-12-07 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation and Flutter
Keywords: New oral anticoagulants; Blood levels; Octogenarians
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample

GROUPS / COHORTS (6):
- octogenarians patients - Apixaban: octogenarians patients who will be treated with Apixaban
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)
- younger than 70 years patients - Apixaba: younger than 70 years patients who will be treated with Apixaba
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)
- octogenarians patients - Rivaroxaban: octogenarians patients who will be treated with Rivaroxaban
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)
- younger than 70 years patients - Rivaroxaban: younger than 70 years patients who will be treated with Rivaroxaban
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)
- octogenarians patients - Dabigatran: octogenarians patients who will be treated with Dabigatran
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)
- younger than 70 years patients - Dabigatran: younger than 70 years patients who will be treated with Dabigatran
  Interventions: Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)

INTERVENTIONS:
Other: New oral anticoagulant pharmacodynamic analysis (blood level assesment)

SUMMARY:
Background: The incidence of atrial fibrillation(AF) increases substantially with age and it is estimated that more than one third of AF patients are octogenarians. Direct oral anticoagulants (DOACs) were found favorable compared to warfarin with respect to efficacy and safety ( bleeding) across wide range of ages.

Nevertheless, the rates of bleeding among elderly patients were shown to increase substantially with all anticoagulants. Dose-adjustments of DOAC are not universally performed among patients older than 80 years old and currently there is paucity of data regarding the actual drugs level among these patients. Accordingly, the investigators sought to investigate the drug levels of the different DOACs among "real world" octogenarians who receiving guideline-recommended dosage.

Methods: A cross sectional, prospective study of 120 hospitalized and ambulatory patients who are treated with DOACs for AF.

DOACs blood levels with be compared between octogenarians (n=70) and younger patient group ( age≤70 year-old; n=50).The cohort will include: 1)Sixty patients on APIXABAN: 40 octogenarians and 20 younger than 70 years, 2)Forty patients on RIVAROXABAN: 20 octogenarians and 20 younger than 70 years, and 3) Twenty patients treated with DABIGATRAN: 10 octogenarians and 10 younger than 70 years.

DOACs Pharmacodynamic analysis will be performed using commercial kits for diluted thrombin time(DTT) and anti-factor Xa activity (AFXa). Drug level will be measured at steady state( through levels) and at Tmax after at least 4 days of complete adherence for DOAC consumption.

Study End-Points:The study main objectives are: 1) DOACs levels in octogenarians in comparison to patients younger than 70 years and 2)percentage of patients, in each group, who have target DTT or AFXa ( predicted) at steady state.

Potential significance of the study:

The results of the study may provide new data on DOACs levels in octogenarians and thus would either support current recommendations or set the ground for further studies aim to optimize DOACs dosage in this vulnerable population.

DETAILED DESCRIPTION:
A cross sectional, prospective study of hospitalized and ambulatory patients, who are treated with DOACs for AF.

Patient population Candidate for the study will be patients older than 80 years (octogenarians) and those ≤70 years who are 1) admitted to the Internal Medicine division in Rabin Medical Center or to Beit Rivka rehabilitation hospital who are on treatment of DOAC prior to their hospitalization \ rehabilitation , 2) hospitalized patients in whom DOAC will be initiated during hospitalization and 3) referred ambulatory patients on DOACs. Each potential patient will be screened for age and other risk factors for bleeding (specifically those that requires dose adjustment such as renal failure, weight, potentially interacting drugs) under DOAC treatment.

Study cohorts

The investigators plan to assess DOACS levels among 120 patients who will be treated by one of the three available agents:

Group 1) sixty patients who will be treated with the direct Xa inhibitor Apixaban - 40 octogenarians and 20 younger than 70 years.

Group 2) forty patients who will be treated with direct Xa inhibitor Rivaroxaban - 20 octogenarians and 20 younger than 70 years Group 3) twenty patients who will be treated with the direct Thrombin inhibitor Dabigatran - 10 octogenarian patients who will receive age-adjusted recommended reduced dosage (110 mg bid) and 10 patients younger than 70 years.

Decision to continue and/or to initiate DOAC as well the dosage, will be on the discretion of the treating physician. Patients in whom the prescribed dosage will not be according to current recommendations will be excluded, unless appropriate adjustment will be made prior to enrolment.

Informed consent will be obtained from all patients prior to study enrolment. Patient's demographic data will be documented at baseline and will include: age, sex, body weight and height, comorbidities, concurrent medications, blood test results (complete blood count, INR, aPTT, renal function tests, electrolytes and liver enzymes). CHA2DS2-VASc and HAS-BLED risk scores will be calculated for each enrolled patient. Actual body weight will be determined upon recruitment with a standardized, calibrated scale.

DOACs pharmacodynamic analysis will be performed using commercial kits for DTT and AFXa. Drug levels will be measured at steady state (through levels) and at Tmax (the time at which maximum serum peak concentration is observed).

DTT and AFXa will be sampled after at least 4 days of complete adherence for DOAC consumption. In the case of hospitalized patient, drug levels will be obtained prior to patients discharge. The steady state sample will be taken just before the morning dose (trough levels). Maximal DTT and AFXa (at Tmax) will be determined by blood sample taken 2 hours after the morning dose with dabigatran and 3 hours with Apixaban/Rivaroxaban.

All blood samples will be drawn when the patient clinical condition is stable and not differ from his/her baseline daily status (including stable kidney functions). In addition, an adherence to the prescribed dosage of the DOAC for at least 4 consecutive days will be assured prior to blood sampling. Accordingly, hospitalized patients may be discharged and invited later to the ward for drug level sampling based on the discretion of the enrolling physician (for example, in the case of questionable adherence in the last 4 days or to allow full recovery from significant change in medical condition).

All blood samples for the study will be drawn by the attending physician. The blood samples (2 tubes of 3 ml each) will be coded and collected in 3.2% citrated tubes for measurement of the pharmacodynamic effects, which will be performed in Beilinson hospital coagulation lab.

The coding system will be based on patients drug treatment. Dabigtran, Rivaroxaban and Apixaban samples will be coded with the first letter in the generic drug name and a running serial number (such as D-1,2,3…).

Immediately after collection, each tube will be transferred to the coagulation lab, inverted to achieve complete mixing and then centrifuged for 10 min at 3000xg. Platelet-poor plasma will then be transferred to a labeled transfer tube and stored at -20°C. The samples will be kept in the coagulation lab freezer for two months after collection. Chromogenic anti Xa assay analysis will be performed on thawed samples using commercial assay (Liquid anti Xa, Instrumentation Laboratory, MA, USA). Diluted thrombin time assay will be performed on the samples using a commercial assay ( Hemoclot Thrombin Inhibitors, Hyphen Biomed, France).

Inclusion criteria:

* Octogenarian group : Age ≥ 80 years.
* Younger age group: Age ≤ 70 years.
* Previous diagnosis of non-valvular atrial fibrillation / flutter or new diagnosis, documented by electrocardiography
* CHA2DS2-VASc score ≥1.
* Hemodynamically stable patients (i.e., without cardiogenic shock or circulatory collapse).
* Receiving DOACs for at least 4 days.
* Stable renal function.

Exclusion criteria:

* Patients who are expected to stop DOACs within the 4-8 days (i.e. planned operation or invasive procedure)
* Patients who require dose adjustment of DOACs based on clinical judgment and not on manufacturer recommendations (i.e. acute renal function deterioration with GFR less than 30 ml/min, need for dual antiplatelet therapy)
* History of gastrointestinal conditions that could significantly impact drug absorption (such as Crohn's disease, gastrectomy).
* A history of recent drug or alcohol abuse
* Concomitant treatment with combined strong P-gp inhibitors and CYP3A4 inhibitors drugs (such as: grapefruit juice, itraconazole, lopinavir/ritonavir, clarithromycin, ritonavir, ketoconazole, indinavir/ritonavir, conivaptan).
* Concomitant treatment with combined strong P-gp inducers and CYP3A4 inducers drugs (such as: avasimibe ,carbamazepine, phenytoin, phenobarbital, rifampin, St John's wort)
* Estimated glomerular filtration rate < 30 ml/min
* Patients with elevated liver enzymes ALT/AST > 3 x ULN or total bilirubin ≥ 1.5 x ULN.
* Weight > 120 kg.
* Pregnant woman.

Study termination criteria:

•None.

Study duration- The study expected duration is 2 years.

Statistical analysis - The sample size for this study was chosen to provide a cohort large enough to identify differences between groups, based on previous studies. Descriptive statistics will be used to calculate summary data. Data will be represented as mean ± SD or as median [5th, 95th percentile], unless otherwise indicated.

Parametric, two-tailed Student's t-tests or ANOVA will be used for continuous variables and the χ2 and Fisher's exact test for categorical variables with a predetermined alpha level of P < 0.05. Statistical analysis will be performed using SAS statistical software (version 8.2, SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Octogenarian group : Age ≥ 80 years.
* Younger age group: Age ≤ 70 years.
* Previous diagnosis of non-valvular atrial fibrillation / flutter or new diagnosis, documented by electrocardiography
* CHA2DS2-VASc score ≥1.
* Hemodynamically stable patients (i.e., without cardiogenic shock or circulatory collapse).
* Receiving DOACs for at least 4 days.
* Stable renal function.

Exclusion Criteria:

* Patients who are expected to stop DOACs within the 4-8 days (i.e. planned operation or invasive procedure)
* Patients who require dose adjustment of DOACs based on clinical judgment and not on manufacturer recommendations (i.e. acute renal function deterioration with GFR less than 30 ml/min, need for dual antiplatelet therapy)
* History of gastrointestinal conditions that could significantly impact drug absorption (such as Crohn's disease, gastrectomy).
* A history of recent drug or alcohol abuse
* Concomitant treatment with combined strong P-gp inhibitors and CYP3A4 inhibitors drugs (such as: grapefruit juice, itraconazole, lopinavir/ritonavir, clarithromycin, ritonavir, ketoconazole, indinavir/ritonavir, conivaptan).
* Concomitant treatment with combined strong P-gp inducers and CYP3A4 inducers drugs (such as: avasimibe ,carbamazepine, phenytoin, phenobarbital, rifampin, St John's wort)
* Estimated glomerular filtration rate < 30 ml/min
* Patients with elevated liver enzymes ALT/AST > 3 x ULN or total bilirubin ≥ 1.5 x ULN.
* Weight > 120 kg.
* Pregnant woman.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Candidate for the study will be patients older than 80 years (octogenarians) and those ≤70 years who are 1) admitted to the Internal Medicine division in Rabin Medical Center or to Beit Rivka rehabilitation hospital who are on treatment of DOAC prior to their hospitalization \ rehabilitation , 2) hospitalized patients in whom DOAC will be initiated during hospitalization and 3) referred ambulatory patients on DOACs. Each potential patient will be screened for age and other risk factors for bleeding (specifically those that requires dose adjustment such as renal failure, weight, potentially interacting drugs) under DOAC treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Diluted thrombin time (DTT) for Dabigatran | trough and peak levels after at least 4 days of drug intake (trough will be taken just before the morning dose and peak levels 2 hours after the intake of Dabigatran)
anti FXa-activity for Apixaban and Rivaroxaban | trough and peak levels after at least 4 days of drug intake (trough will be taken just before the morning dose and peak levels 3 hours after the intake of Apixaba/Rivaroxaban)

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Fuches, MD, Study Chair — Internal Medicine B Department, Rabin Medical Center, Beilinson Hospital; Ran Nissan, PharmD, Principal Investigator — Internal Medicine B Department, Rabin Medical Center, Beilinson Hospital; Shai Shimoni, MD, Principal Investigator — Internal Medicine B Department, Rabin Medical Center, Beilinson Hospital
Locations (2):
- Israel (2):
  - Internal Medicine B Department, Petah Tikva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva

REFERENCES:
- [Background] Haim M, Hoshen M, Reges O, Rabi Y, Balicer R, Leibowitz M. Prospective national study of the prevalence, incidence, management and outcome of a large contemporary cohort of patients with incident non-valvular atrial fibrillation. J Am Heart Assoc. 2015 Jan 21;4(1):e001486. doi: 10.1161/JAHA.114.001486. PMID 25609415
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines-CPG; Document Reviewers. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation--developed with the special contribution of the European Heart Rhythm Association. Europace. 2012 Oct;14(10):1385-413. doi: 10.1093/europace/eus305. Epub 2012 Aug 24. No abstract available. PMID 22923145
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Miller CS, Grandi SM, Shimony A, Filion KB, Eisenberg MJ. Meta-analysis of efficacy and safety of new oral anticoagulants (dabigatran, rivaroxaban, apixaban) versus warfarin in patients with atrial fibrillation. Am J Cardiol. 2012 Aug 1;110(3):453-60. doi: 10.1016/j.amjcard.2012.03.049. Epub 2012 Apr 24. PMID 22537354
- [Background] Sardar P, Chatterjee S, Chaudhari S, Lip GY. New oral anticoagulants in elderly adults: evidence from a meta-analysis of randomized trials. J Am Geriatr Soc. 2014 May;62(5):857-64. doi: 10.1111/jgs.12799. Epub 2014 May 1. PMID 24786913
- [Background] Halvorsen S, Atar D, Yang H, De Caterina R, Erol C, Garcia D, Granger CB, Hanna M, Held C, Husted S, Hylek EM, Jansky P, Lopes RD, Ruzyllo W, Thomas L, Wallentin L. Efficacy and safety of apixaban compared with warfarin according to age for stroke prevention in atrial fibrillation: observations from the ARISTOTLE trial. Eur Heart J. 2014 Jul 21;35(28):1864-72. doi: 10.1093/eurheartj/ehu046. Epub 2014 Feb 20. PMID 24561548
- [Background] Held C, Hylek EM, Alexander JH, Hanna M, Lopes RD, Wojdyla DM, Thomas L, Al-Khalidi H, Alings M, Xavier D, Ansell J, Goto S, Ruzyllo W, Rosenqvist M, Verheugt FW, Zhu J, Granger CB, Wallentin L. Clinical outcomes and management associated with major bleeding in patients with atrial fibrillation treated with apixaban or warfarin: insights from the ARISTOTLE trial. Eur Heart J. 2015 May 21;36(20):1264-72. doi: 10.1093/eurheartj/ehu463. Epub 2014 Dec 12. PMID 25499871
- [Background] Stollberger C, Finsterer J. Concerns about the use of new oral anticoagulants for stroke prevention in elderly patients with atrial fibrillation. Drugs Aging. 2013 Dec;30(12):949-58. doi: 10.1007/s40266-013-0119-3. PMID 24170233
- [Derived] Nissan R, Spectre G, Hershkovitz A, Green H, Shimony S, Cooper L, Nakav S, Shochat T, Grossman A, Fuchs S. Apixaban Levels in Octogenarian Patients with Non-valvular Atrial Fibrillation. Drugs Aging. 2019 Feb;36(2):165-177. doi: 10.1007/s40266-018-0613-8. PMID 30460518